CLINICAL TRIAL: NCT01857518
Title: Depression in Adolescents. A Cerebral Structural, Diffusion, and Functional Magnetic Resonance Imaging Study.
Acronym: ADODEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier St Anne (Other)
Collaborators: CENIR Centre de Neuroimagerie de Recherche, Paris (Unknown); Inserm CEA Research unit U1000 (Neuroimaging in psychiatry) (Unknown); National Research Agency, France (Other); Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 2012-A01466-37; D500 (Other: CHSA)
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Adolescent Depression
MeSH Terms: interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Depressed adolescents Group (Other): Adolescents with a major depressive episode diagnosis
  Interventions: Other: -Diagnostic, clinical and psycho-behavioral assessments -Neuroimaging: T1-MRI, DTI-MRI, fMRI
- Healthy adolescent control Group (Other): Healthy adolescents recruited from general population
  Interventions: Other: -Diagnostic, clinical and psycho-behavioral assessments -Neuroimaging: T1-MRI, DTI-MRI, fMRI

INTERVENTIONS:
Other: -Diagnostic, clinical and psycho-behavioral assessments -Neuroimaging: T1-MRI, DTI-MRI, fMRI — * Visit V1: Diagnostic and clinical assessments
  * Visit V2: psycho-behavioral assessment and neuroimaging
  * Visit V3: Diagnostic and clinical assessments
  * Visit V4: psycho-behavioral assessment and neuroimaging

SUMMARY:
Adolescence is a critical period for the development of depressive disorders. As adolescence also is a critical period for brain maturation, it may be hypothesized that maturation changes in emotional circuits could underlie vulnerability for depression.

The aims of the study are (1) to identify the changes in brain morphometry, white matter microstructure, and functioning, in networks associated with depression features in adolescents, and (2) to assess the effects of treated pathology on brain structure by comparing the neuroimaging measures obtained in adolescents at inclusion with those at follow-up.

DETAILED DESCRIPTION:
Adolescence is a key development period for neurobiological processes underlying emotional and cognitive functions in adulthood. The pathophysiology of mood disorders has recently been associated with maturation changes in brain networks, but little is known on the early brain structure changes associated with depression appearing during this major brain maturation period.

The hypothesis of altered structural integrity of limbic prefrontal pathways emerges from the literature on depression, but it is unknown whether it is also detectable in adolescents with depression. Thus, we aim to investigate WM and GM structure and anatomy, and functional correlates of behavioral responses in depressed adolescents.

40 adolescents with a Major Depressive Episode will be investigated using structural T1 magnetic-resonance imaging and diffusion tensor imaging (DTI), at inclusion and after one-year follow-up. Additionally, they will be investigated with fMRI.

Covariation patterns between neuroimaging and behavioural/clinical variables will be assessed.

ELIGIBILITY:
Inclusion Criteria:

Depressed adolescents:

Teenagers of both sexes, from 15 to 18 years old, without contreindications in magnetic fields

* affiliation to a Social insurance
* Informed consent signed by the holders of the parental rights (a specific information note to the teenager)
* Diagnosis DSM-IV-TR ( 2000 ) of depressive Disorder of the humor without psychotic characteristics. The symptoms will have to be persistent for 3 weeks, in spite of a coverage of support ( 2 consultations).

Exclusion Criteria:

* Ferromagnetical Material in the body
* Claustrophobia, Syndrom of post-traumatic stress, Obsessive-compulsive Disorder, Disturb Tricks, Disturbs abuse of substances
* Intrusive disorder of the development, Disturbs hyperactivity deficit of the attention, Disorders of the conducts, Schizophrenia
* Current antidepressant or antipsychotic psychotropic Treatment for more than 15 days in effective doses
* Current somatic pathology, or pregnancy (urinary test of pregnancy in case of doubt)
* Histories of cranial trauma or neurological pathology, or of lower born weight in 800g
* History of electroconvulsivotherapy in the previous 6 months
* Refusal to give his(her) consent or to be revised on one year after inclusion

Healthy adolescents: will be screened to be matched to the patients according to age and sex. They will have no psychiatric diagnosis, and no family history of psychiatric conditions.

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-08-31 (Actual); Primary Completion 2018-02 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Evidence of white matter microstructure changes | Baseline
  Statistical map of voxel-based analysis of white matter using tract based spatial statistics (TBSS) to compare depressed adolescents and healthy controls in emotional and reward networks
Evidence of grey matter volume changes | Baseline
  Statistical map of voxel-based analysis of grey matter using statistical parametric mapping (SPM8) to compare depressed adolescents and healthy controls in emotional and reward networks

SECONDARY OUTCOMES:
Correlation between Functional anatomy of emotional/reward responses and white matter and grey matter structure changes | Baseline
Grey matter and white matter changes in frontal limbic networks at follow-up in treated patients | Follow-up one year

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Laure PAILLERE MARTINOT, MD, PhD, Principal Investigator — APHP
Locations (1):
- Cochin Hospital, Paris, France